CLINICAL TRIAL: NCT05883956
Title: A Phase 3b, Randomized, Open-Label, Double Crossover Study Comparing Treatment Preference Between Oral Decitabine/Cedazuridine and Azacitidine in Adult Patients With IPSS R Intermediate Myelodysplastic Syndrome, Low Blast Acute Myeloid Leukemia, IPSS Intermediate-2 or High Risk Myelodysplastic Syndrome or Chronic Myelomonocytic Leukemia
Brief Title: A Study Comparing Treatment Preference Between Oral Decitabine/Cedazuridine and Azacitidine in Myelodysplastic Syndrome, Low-Blast Acute Myeloid Leukemia, or Chronic Myelomonocytic Leukemia
Acronym: PREFER-HMA
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Australia Pharmaceutical Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 393-419-00041
Record Dates: First submitted 2023-04-25; First posted 2023-06-01 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Myelodysplastic Syndromes; Leukemia, Myeloid, Acute; Leukemia, Myelomonocytic, Chronic; Patient Preference
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myeloid, Acute; Leukemia, Myelomonocytic, Chronic; Patient Preference | interventions — decitabine and cedazuridine drug combination

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ABBA (Active Comparator): Cycle 1: Oral decitabine/cedazuridine; Cycle 2: Subcutaneous azacitidine; Cycle 3: Subcutaneous azacitidine; Cycle 4: Oral decitabine/cedazuridine
  Interventions: Drug: Subcutaneous azacitidine; Drug: Oral decitabine/cedazuridine
- BAAB (Active Comparator): Cycle 1: Subcutaneous azacitidine; Cycle 2: Oral decitabine/cedazuridine; Cycle 3: Oral decitabine/cedazuridine; Cycle 4: Subcutaneous azacitidine
  Interventions: Drug: Subcutaneous azacitidine; Drug: Oral decitabine/cedazuridine

INTERVENTIONS:
Drug: Subcutaneous azacitidine — Subcutaneous azacitidine, 75mg/m2, 7 days
Drug: Oral decitabine/cedazuridine — Oral decitabine 35mg/cedazuridine 100mg, once daily, 5 days

SUMMARY:
It is hypothesized that significantly more patients would prefer oral decitabine/cedazuridine to subcutaneous (SC) azacitidine (AZA) due to several factors, including improved treatment convenience, the reduced risk of nosocomial infections, and reduced treatment discomfort. However, this hypothesis has not been formally studied in a controlled setting. This study aims to address this evidence gap and evaluate patient, primary caregiver (carer), and clinician treatment preference between oral decitabine/cedazuridine and SC AZA in the treatment of adult patients with International Prognostic Scoring System-Revised (IPSS-R) intermediate, IPSS intermediate-2, or high-risk myelodysplastic syndrome (MDS), chronic myelomonocytic leukemia (CMML), or low-blast (LB) acute myeloid leukemia (AML) and thereby lend further credibility to the clinical, economic, and patient value of oral decitabine/cedazuridine.

ELIGIBILITY:
Inclusion Criteria:

For Patients:

Patients are eligible to be included in the study only if all of the following criteria apply at any time starting from Screening up to Day 1 prior to study treatment administration:

* Patients must be 18 years of age or older.
* IPSS-R defined intermediate MDS, IPSS defined intermediate 2 or high-risk MDS, LB AML or CMML (with symptoms), as confirmed by recent full blood examination, bone marrow biopsy, and cytogenetic testing. NOTE: IPSS-R defined intermediate MDS patients are limited to less than 50% of enrolled patients.
* Life expectancy of at least 6 months.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 2 inclusive.
* Patient must be able to co-operate and complete tasks (including tasks such as electronic questionnaires on digital devices) over the following 4 months.

Inclusion Criteria:

For Patients:

Patients are eligible to be included in the study only if all of the following criteria apply at any time starting from Screening up to Day 1 prior to study treatment administration:

* Patients must be 18 years of age or older.
* IPSS-R defined intermediate MDS, IPSS defined intermediate 2 or high-risk MDS, LB AML or CMML (with symptoms), as confirmed by recent full blood examination, bone marrow biopsy, and cytogenetic testing. NOTE: IPSS-R defined intermediate MDS patients are limited to less than 50% of enrolled patients.
* Life expectancy of at least 6 months.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 2 inclusive.
* Patient must be able to co-operate and complete tasks (including tasks such as electronic questionnaires on digital devices) over the following 4 months.
* Patient must be able to identify a carer to participate in completing the cTPMQ.

For Carers:

• Primary carer of a patient meeting all of the inclusion criteria (ie, a patient who meets criteria defined above).

For Clinicians:

• Clinician treating patients meeting all of the inclusion criteria (ie, treats patients who meet criteria defined above).

Exclusion Criteria:

For Patients:

Patients are excluded from the study if any of the following criteria apply:

* Patients with known hypersensitivity to the study treatments oral decitabine/cedazuridine or azacitidine.
* Patients with advanced malignant hepatic tumors.
* Patients with severe renal impairment (creatinine clearance <30 mL/min).
* Patients who have received hypomethylating agents (HMA) previously.
* Patients who are receiving lenalidomide or are receiving other therapies outside of standard of care (SOC).
* Receipt of any immunotherapy, any conventional or investigational systemic anti-cancer therapy within 5 half-lives of the drug, or within 4 weeks prior to the first dose of study treatment (whichever is longer).
* Any medical, psychological, social, or other condition which in the view of the Investigator is likely to interfere with the study, compliance, or put the patient at risk.
* Participants who are not fluent in English, or who cannot read or write in English will be excluded from the study.

For Carers:

Carers are excluded from the study if any of the following criteria apply:

* They are a carer of a patient who meets any of the exclusion criteria listed above.
* They are a relative of an employee of the investigational clinic or sponsor (e.g. Investigator, study coordinator)

For Clinicians:

• Clinicians will be excluded from participating in the study if they are a relative of an employee of the investigational clinic or sponsor (e.g. Investigator, Study Coordinator).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2023-12-20 (Actual); Primary Completion 2024-12-06 (Actual); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients reporting preference for oral decitabine/cedazuridine vs subcutaneous azacitidine on the patient treatment preference in myelodysplasia questionnaire (pTPMQ) | Prior to initiation of Cycle 3 (each cycle is 28 days)
Proportion of patients reporting preference for oral decitabine/cedazuridine vs subcutaneous azacitidine on the pTPMQ | Prior to initiation of Cycle 5 (each cycle is 28 days)

SECONDARY OUTCOMES:
Proportion of carers reporting preference for oral decitabine/cedazuridine vs subcutaneous azacitidine on the carer treatment preference in myelodysplasia questionnaire (cTPMQ) | Prior to initiation of Cycle 3 (each cycle is 28 days)
Proportion of carers reporting preference for oral decitabine/cedazuridine vs subcutaneous azacitidine on the cTPMQ | Prior to initiation of Cycle 5 (each cycle is 28 days)
Proportion of clinicians reporting preference for oral decitabine/cedazuridine vs subcutaneous azacitidine on the medical treatment preference in myelodysplasia questionnaire (mTPMQ) | Prior to initiation of Cycle 4 (each cycle is 28 days)
Proportion of clinicians reporting preference for oral decitabine/cedazuridine vs subcutaneous azacitidine on the mTPMQ | End of Study (EOS) Day 28
Proportion of clinicians choosing oral decitabine/cedazuridine vs subcutaneous azacitidine for continuation of treatment and reasons for the treatment choice based on the mTPMQ | Cycle 5, Day 1 (each cycle is 28 days)
Difference in quality of life between oral decitabine/cedazuridine and subcutaneous azacitidine as assessed using the EQ-5D-5L in Myelodysplastic Syndrome, Chronic Myelomonocytic Leukemia and Low-Blast Acute Myeloid Leukemia patients | Cycle 1, Day 1 (each cycle is 28 days)
Difference in quality of life between oral decitabine/cedazuridine and subcutaneous azacitidine as assessed using the EORTC QLQ-C30 in Myelodysplastic Syndrome, Chronic Myelomonocytic Leukemia and Low-Blast Acute Myeloid Leukemia patients | Cycle 1, Day 1 (each cycle is 28 days)
Difference in quality of life between oral decitabine/cedazuridine and subcutaneous azacitidine as assessed using the EQ-5D-5L in Myelodysplastic Syndrome, Chronic Myelomonocytic Leukemia and Low-Blast Acute Myeloid Leukemia patients | Cycle 3, Day 5 (each cycle is 28 days)
Difference in quality of life between oral decitabine/cedazuridine and subcutaneous azacitidine as assessed using the EORTC QLQ-C30 in Myelodysplastic Syndrome, Chronic Myelomonocytic Leukemia and Low-Blast Acute Myeloid Leukemia patients | Cycle 3, Day 5 (each cycle is 28 days)
Difference in quality of life between oral decitabine/cedazuridine and Subcutaneous azacitidine as assessed using the EQ-5D-5L in Myelodysplastic Syndrome, Chronic Myelomonocytic Leukemia and Low-Blast Acute Myeloid Leukemia patients | Cycle 4, Day 5 (each cycle is 28 days)
Difference in quality of life between oral decitabine/cedazuridine and Subcutaneous azacitidine as assessed using the EORTC QLQ-C30 in Myelodysplastic Syndrome, Chronic Myelomonocytic Leukemia and Low-Blast Acute Myeloid Leukemia patients | Cycle 4, Day 5 (each cycle is 28 days)
Difference in quality of life between oral decitabine/cedazuridine and subcutaneous azacitidine as assessed using the EQ-5D-5L in Myelodysplastic Syndrome, Chronic Myelomonocytic Leukemia and Low-Blast Acute Myeloid Leukemia patients | Cycle 5, Day 5 (each cycle is 28 days)
Difference in quality of life between oral decitabine/cedazuridine and subcutaneous azacitidine as assessed using the EORTC QLQ-C30 in Myelodysplastic Syndrome, Chronic Myelomonocytic Leukemia and Low-Blast Acute Myeloid Leukemia patients | Cycle 5, Day 5 (each cycle is 28 days)
Difference in quality of life between oral decitabine/cedazuridine and subcutaneous azacitidine as assessed using the EQ-5D-5L in Myelodysplastic Syndrome, Chronic Myelomonocytic Leukemia and Low-Blast Acute Myeloid Leukemia patients | Cycle 6, Day 5 (each cycle is 28 days)
Difference in quality of life between oral decitabine/cedazuridine and subcutaneous azacitidine as assessed using the EORTC QLQ-C30 in Myelodysplastic Syndrome, Chronic Myelomonocytic Leukemia and Low-Blast Acute Myeloid Leukemia patients | Cycle 6, Day 5 (each cycle is 28 days)
The difference in the incidence of treatment discontinuation and reasons for treatment discontinuation | Baseline (pre-intervention) through to study completion (up to 6 cycles of treatment where each cycle is 28 days)
Incidence and severity of adverse events upon study physician discretion. | Baseline (pre-intervention) through to study completion (up to 6 cycles of treatment where each cycle is 28 days)

CONTACTS AND LOCATIONS:
Overall Officials: Anoop Enjeti, Principal Investigator — Calvary Mater Newcastle, Edith Street, Waratah, NSW 2298 Australia
Locations (11):
- Australia (6):
  - Calvary Mater Newcastle, Newcastle, New South Wales
  - Pindara Private Hospital, Benowa, Queensland
  - Townsville Hospital, Townsville, Queensland
  - Adelaide Oncology and Haematology, North Adelaide, South Australia
  - Grampian Health (Ballarat Base Hospital), Ballarat Central, Victoria
  - Latrobe Regional Hospital, Traralgon, Victoria
- New Zealand (5):
  - Christchurch Hospital, Christchurch
  - Dunedin Hospital, Dunedin
  - Auckland City Hospital, Grafton
  - Waikato Hospital, Hamilton
  - North Shore Hospital (Waitemata District Health Board), Takapuna

IPD SHARING:
Plan to Share IPD: No